CLINICAL TRIAL: NCT02113514
Title: Community Awareness, Resources and Education (CARE I): Project 3
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-0490
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Abnormality
Keywords: Appalachian; abnormal pap test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cervical mucus will be collected for Human Papillomavirus (HPV) assays and stored for potential other assays related to HPV. Serum will be drawn for HPV serology and stored for future analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal Pap smear: Women with normal pap test.
- Abnormal Pap smear: Women with abnormal pap test.

SUMMARY:
Community Awareness, Resources and Education (CARE) Project - Project 3 will determine if Appalachian women have unique risk factors for an abnormal Pap smear that might contribute to the increased risk of cervical abnormalities, specifically cancer, in their communities.

DETAILED DESCRIPTION:
The aim of CARE: Project 3 is to determine the social, behavioral, and biological variables that might contribute to increased risks of an abnormal Pap smear in Appalachian women in Ohio. To accomplish these aims, a case-control study was proposed. Women age 18 and older with an intact cervix, not pregnant, and no current or past history of invasive cervical cancer are recruited at the time of their scheduled Pap smear from clinics/physician practices in Appalachian region of Ohio. Women receiving Pap tests at participating medical clinics/physician practices are recruited for a case control epidemiologic study assessing HPV prevalence and its impact on cervical intraepithelial neoplasia (CIN). Cervical mucus will be collected for Human Papillomavirus (HPV) assays and stored for potential other assays related to HPV. Serum will be drawn for HPV serology and stored for future analysis. Controls are defined as women with a normal Pap smear. Cases are defined as women with abnormal Pap smear (from atypical squamous cells of uncertain significance (ASCUS) to cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years or older
* Able to give informed consent
* Intact cervix
* No prior history of invasive cervical cancer
* English speaking
* Willing to have biological specimens stored for future studies
* Resident of Appalachian Ohio

Exclusion Criteria:

* Pregnant
* Medical or psychiatric illness that precludes research project requirements, ability to give informed consent, or protocol compliance.
* Smokers (will be contacted by study team to see if they are eligible/willing to participate in CARE: Project 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Woman 18 years or older that are nonpregnant with intact cervix and no cervical cancer who present for a Pap smear. Must be residents of an Appalacian Ohio county.
Sampling Method: Non-Probability Sample
Enrollment: 2394 (Actual)
Dates: Start 2005-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Social/environmental variables of access to screening were analyzed to see if they contribute to increased risk of developing abnormalities among Appalachian women. | Participant completed all activites on the 1 day of the clinic visit.
  On the day of study enrollment, survey data and specimens were obtained from the participants.

SECONDARY OUTCOMES:
Behavioral variables of age of onset of sexual intercourse, number of partners, male partner factors, multiparity, oral contraceptive use, and smoking were analyzed to see if they contribute to the increased risk of developing abnormalities. | Participant completed all activites on the 1 day of the clinic visit.
  On the day of study enrollment, survey data and specimens were obtained from the participants.
Biological variables of HPV status, HPV type, HPV variants, HPV viral load, and serology to HPV were analyzed to see if they contribute to the increased risk of developing cervical abnormalities among Appalachian women. | Participant completed all activites on the 1 day of the clinic visit.
  On the day of study enrollment, survey data and specimens were obtained from the participants.
Combinations of social, behavioral, and biological determinants were analyzed to see which contribute to the increased risk of developing cervical abnormalities among Appalachian women. | Participant completed all activites on the 1 day of the clinic visit.
  On the day of study enrollment, survey data and specimens were obtained from the participants.

OTHER OUTCOMES:
Factors that impede follow-up and treatment of abnormal or suspicious Pap smear findings were identified. | Participant completed all activites on the 1 day of the clinic visit.
  On the day of study enrollment, survey data and specimens were obtained from the participants.
New molecular markers related to cervical cancer were explored. | Participant completed all activites on the 1 day of the clinic visit.
  On the day of study enrollment, survey data and specimens were obtained from the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D. Paskett, PhD, Principal Investigator — The Ohio State University Center for Population Health and Health Disparities
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - The Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Patel DA, Rozek LS, Colacino JA, Van Zomeren-Dohm A, Ruffin MT, Unger ER, Dolinoy DC, Swan DC, Onyekwuluje J, DeGraffinreid CR, Paskett ED. Patterns of cellular and HPV 16 methylation as biomarkers for cervical neoplasia. J Virol Methods. 2012 Sep;184(1-2):84-92. doi: 10.1016/j.jviromet.2012.05.022. Epub 2012 Jun 1. PMID 22664184
- [Result] Ruffin MT 4th, Hade EM, Gorsline MR, DeGraffinreid CR, Katz ML, Kobrin SC, Paskett ED. Human papillomavirus vaccine knowledge and hypothetical acceptance among women in Appalachia Ohio. Vaccine. 2012 Aug 3;30(36):5349-57. doi: 10.1016/j.vaccine.2012.06.034. Epub 2012 Jun 27. PMID 22749839
- [Result] Reiter PL, Katz ML, Ruffin MT, Hade EM, DeGraffenreid CR, Patel DA, Paskett ED, Unger ER. HPV prevalence among women from Appalachia: results from the CARE project. PLoS One. 2013 Aug 30;8(8):e74276. doi: 10.1371/journal.pone.0074276. eCollection 2013. PMID 24023700
- See also: Jamesline — http://cancer.osu.edu